CLINICAL TRIAL: NCT07028463
Title: ALERT-ED: Awareness and Linkage to Resources for At-Risk Emergency Department Patients
Acronym: ALERT-ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-1263
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: High Fall Risk
Keywords: Fall risk; Automated notification; resource referral; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receives online educational recourses (No Intervention)
- ALERT-ED (Experimental): Patient receives link to the Livi Chatbot in After Visit Summary
  Interventions: Behavioral: ALERT-ED

INTERVENTIONS:
Behavioral: ALERT-ED — Patient receives link to the Livi Chatbot in After Visit Summary
  Arms: ALERT-ED

SUMMARY:
Falls are the leading reason for injury-related emergency department (ED) visits in older adults with high rates of ED revisits for falls. Evidence-based fall prevention programs can reduce falls by 30%, but older adults commonly describe limited awareness of resources. Currently, all UCHealth ED patients receive fall risk screening on ED arrival, but patients are rarely made aware of their screening results or referred to resources. To address this gap, our team developed ALERT-ED, an intervention where study patients receive automated notification of fall risk screening results and referral via Livi to evidence-based fall prevention programs near their homes. If ALERT-ED is successful, we will demonstrate that UCHealth can improve patient health via pragmatic, automated notification of screening results and referral to resources. Although we designed ALERT-ED to intervene on fall risk in EDs, the intervention could be used for other health concerns central to UCHealth's mission including for patients seeking care for transplants, cancer, brain health, or orthopedic concerns.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Screens high risk falls on the Geriatric Fall assessment tool (as shown in protocol and used as standard practice in study ED)

Exclusion Criteria:

* Does not consent to follow up interview

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20700 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of fall-related ED visits | 6 months

SECONDARY OUTCOMES:
Patient reported engagement with community fall prevention programs | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UCHealth, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No